CLINICAL TRIAL: NCT00373802
Title: A Randomized, Double-Blinded Placebo Control Trial of Nasal Phenylephrine in Infants With Bronchiolitis
Brief Title: The Use of Nasal Phenylephrine in Infants With Bronchiolitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Nathan Kraynack, M.D., Akron Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NASAL #9579
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine

SUMMARY:
Drops of either saline or phenylephrine are placed in the nose of infants less than 12 months of age to determine if it helps them to breathe easier.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 weeks to 12 months; admitting diagnosis of bronchiolitis; admitted to hospital's bronchiolitis pathway, admitted during weekdays, need for nasal suctioning.

Exclusion Criteria:

* Congenital heart disease, history of hypertension, previous wheezing, prior use of inhaled corticosteroids, gestational age at birth of <34 weeks.

Ages: 4 Weeks to 12 Months | Sex: All
Age Groups: Child
Enrollment: 50
Dates: Start 2005-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Respiratory Distress Assessment Index at 5 minutes, 60 minutes, and 180 minutes.

SECONDARY OUTCOMES:
Respiratory rate, oxygen saturation and use of supplemental oxygen at 5, 60, and 180 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Konda-Sundheim, MD, MD, Principal Investigator — Children's Hospital Medical Center of Akron